CLINICAL TRIAL: NCT03626987
Title: Identification of Protein Markers of Epidemiological and Clinical Interest by MALDI-TOF
Acronym: SPECTRASURV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-16; TPS 15219ter (Registry Identifier: INDS number)
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Infectious Risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bacterial identification: Describe the MALDI-TOF spectrum to identify peaks that may be associated with epidemiological and clinical characteristics of bacterial strains
  Interventions: Diagnostic Test: mass spectrometry (MALDI-TOF)

INTERVENTIONS:
Diagnostic Test: mass spectrometry (MALDI-TOF) — The determination of the protein composition of the bacterial spectrum

SUMMARY:
Not all infectious agents have the same epidemic potential, and this can vary widely within the same species. Rapid determination of this potential is essential to optimize control of infectious diseases. It is now accepted that identification with the species is clearly insufficient to identify an epidemic and to carry out epidemiological analyzes. Indeed, if the same bacterial species can present a great diversity of strains, it is organized in clonal complexes having strong variations of clinical and epidemiological expression.

More specifically, on a bio-epidemiological level, the clonal identification of the bacterial agent is a real asset because it can make it possible to identify the highly virulent strains or known to be resistant, the clones associated with nosocomial infections, the source of the infection. an epidemic and to follow its spatio-temporal extension, to know the epidemiological antiquity of the clone, to follow or rebuild a chain of transmission, to discover epidemic clusters.

There are rapid identification techniques, for example by polymerase chain reaction (PCR), but which are targeted at particular genomic compositions previously identified.

Routine bacterial identification now rests on the determination of the protein composition by mass spectrometry (MALDI-TOF). The bacterial spectrum is compared to a reference library of protein composition, thus obtaining an identification equivalent to that based on the 16s RNA (ribonucleic acid 16s) and can descend to an infra-species level.

The aim of this work is to use the proteome part of the MALDI-TOF spectrum to identify peaks that signal clonality and to determine proteomic fingerprintings that can be used for epidemiological and clinical purposes.

Instead of relying on expensive genomic methods, the identification of the clonal characteristics of the strains will rely on the bacterial proteome present on the MALDI-TOF spectrum that is produced during the routine identification of the bacterium.

The results are intended to feed a complementary knowledge base

ELIGIBILITY:
Inclusion Criteria:

* bacterial identification by Matrix Assisted Laser Desorption Ionisation - Time of Flight (MALDI-TOF)

Exclusion Criteria:

* Unidentified strain or noisy spectrum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bacterial identification of patients taken as part of the care
Sampling Method: Probability Sample
Enrollment: 600000 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Ability to find protein peaks that mark epidemic clones | 36 months
  Ability to find protein peaks that mark epidemic clones Association of these clones with epidemic characteristics (age, antibacterial resistance, virulence)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giraud-Gatineau A, Texier G, Fournier PE, Raoult D, Chaudet H. Using MALDI-TOF spectra in epidemiological surveillance for the detection of bacterial subgroups with a possible epidemic potential. BMC Infect Dis. 2021 Oct 28;21(1):1109. doi: 10.1186/s12879-021-06803-3. PMID 34711189